CLINICAL TRIAL: NCT00841867
Title: A Pilot Study Investigating the Effects of Partial Pancreatectomy on Glucose Tolerance
Brief Title: The Role of Pulsatile Insulin Secretion (A Study Investigating the Effects of Partial Pacreatectomy on Glucose Metabolism)
Acronym: Pilot OGTT
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: DK61539; R01DK061539 (NIH)
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Impaired Glucose Tolerance
Keywords: Impaired Glucose Tolerance; Diabetes
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Subjects 18-80 years of age who have previously undergone partial pancreatectomy due to a benign lesion
  Interventions: Procedure: All subjects will undergo a 120 minute Oral Glucose Tolerance Test at study visit 2.
- 2: Healthy control subjects, 18-80 years of age, who have not had partial pancreatectomy.
  Interventions: Procedure: All subjects will undergo a 120 minute Oral Glucose Tolerance Test at study visit 2.

INTERVENTIONS:
Procedure: All subjects will undergo a 120 minute Oral Glucose Tolerance Test at study visit 2. — All subjects will ingest a 75 g glucose solution (Glucola brand) and have blood drawn at 7 timepoints over 120 minutes.

SUMMARY:
The purpose of this study is to examine changes in sugar metabolism that may occur in subjects who have previously had part of their pancreas removed due to a benign lesion.

DETAILED DESCRIPTION:
Beta cells of the pancreas are the insulin producing cells. People with impaired fasting glucose have a beta cell mass ~50% of that of normal glucose tolerant subjects.

A 2006 canine study by Dr. Peter Butler's group at UCLA demonstrated that glucose stimulated insulin secretion was deficient after 50% decrease in beta cell mass after distal pancreatectomy compared to those dogs who had sham surgery. The pancreatectomized dogs had impaired fasting glucose with impaired insulin secretion and insulin resistance. The decreased insulin secretion was a result of decreased insulin secretory pulses or bursts with no change seen in pulse frequency, the same pattern seen in humans with Type 2 diabetes. Conclusions derived from this study include the following:

1. When beta cell mass declines to ~50% the capacity for the remaining beta cells to secrete insulin in appropriate secretory bursts is compromised, leading to a deficit in insulin secretion most obvious on glucose stimulation.
2. The decreased insulin burst mass results in an additional component of insulin resistance, and this together with the compromised capacity for insulin secretion leads to decompensation of glucose regulation and diabetes onset.

How does this translate in humans who have had partial pancreatectomy? In 1990, Kendall and colleagues published a study looking at the effects of hemipancreatectomy in healthy human subjects on insulin secretion and glucose tolerance. These subjects were donors for pancreatic transplantation. They showed that fasting insulin and c-peptide levels were lower one year after hemipancreatectomy. Seven of the 28 donors had abnormal glucose tolerance one year after hemipancreatectomy, but all 28 had normal fasting plasma glucose levels. This study and others like it confirm the development of impaired glucose tolerance after partial pancreatectomy, but pulsatile insulin secretion and hepatic insulin clearance were not measured.

As stated above, the main objective of this pilot study is to establish and quantify the impact of a deficit in beta cell mass, due to partial pancreatectomy for benign tumors, on glucose tolerance. Results of this study may be used to develop a future metabolic study that uses glucose isotopes to establish the effects of partial pancreatectomy on glucose tolerance, basal and stimulated insulin secretion as well as hepatic and extrahepatic insulin sensitivity under conditions of usual physiology. This will enable us to further understand the relationship between loss of beta cells, decreased insulin secretion and increased insulin resistance in humans.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female subjects
* 18-80 years of age who have had
* partial pancreatectomy due to a benign lesion
* OR are healthy control subjects
* are willing to fast (nothing to eat or drink for 10 hours)prior to visits

Exclusion Criteria:

* Pancreatic malignancy
* Chronic pancreatitis
* Pregnant
* On steroid medications such as prednisone

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects 18-80 years of age who have had partial pancreatectomy for benign lesions and healthy controls who have not had pancreas surgery.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2008-12; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
To determine differences in glucose metabolism between subjects who have had partial pancreatectomy due to a benign lesion and those who have not had such a surgery. | Outcome will be determined after all data has been collected.

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA General Clinical Research Center (GCRC), Los Angeles, California, United States